CLINICAL TRIAL: NCT03310008
Title: An Open-label, Phase I Study to Assess the Safety and Clinical Activity of Multiple Doses of NKR-2, Administered Concurrently With the Neoadjuvant FOLFOX Treatment in Patients With Potentially Resectable Liver Metastases From Colorectal Cancer
Brief Title: Dose Escalation and Dose Expansion Phase I Study to Assess the Safety and Clinical Activity of Multiple Doses of NKR-2 Administered Concurrently With FOLFOX in Colorectal Cancer With Potentially Resectable Liver Metastases
Acronym: SHRINK
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Celyad Oncology SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYAD-N2T-003
Record Dates: First submitted 2017-08-02; First posted 2017-10-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Colon Cancer Liver Metastasis

STUDY DESIGN:
Intervention Model Description: Biological: NKR-2 cells The intervention will consist of an infusion of NKR-2 cells administered concurrently to a standard chemotherapy every 2 weeks (14 days) for a total of 3 infusions within 4 weeks (28 days).
  Other Name: NKG2D CAR-T cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose level 1 (escalation (Experimental): The dose escalation arm will use a 3+3 design to determine the maximum tolerated dose.
  Interventions: Biological: NKR-2 cells
- Dose level 2 (escalation) (Experimental): The dose escalation arm will use a 3+3 design to determine the maximum tolerated dose.
  Interventions: Biological: NKR-2 cells
- Dose level 3 (escalation) (Experimental): The dose escalation arm will use a 3+3 design to determine the maximum tolerated dose.
  Interventions: Biological: NKR-2 cells
- Recommended dose level (expansion) (Experimental): The dose expansion arm will use the maximum tolerated dose.
  Interventions: Biological: NKR-2 cells

INTERVENTIONS:
Biological: NKR-2 cells — The intervention will consist of an infusion of NKR-2 cells administered concurrently to a standard chemotherapy every 2 weeks (14 days) for a total of 3 infusions within 4 weeks (28 days).
  Other Names: NKG2D CAR-T cells

SUMMARY:
SHRINK (Standard cHemotherapy Regimen and Immunotherapy with NKR-2) is an open-label Phase I study to assess the safety and clinical activity of multiple administrations of autologous NKR-2 cells administered concurrently with a standard chemotherapy treatment (FOLFOX) in potentially resectable liver metastases from colorectal cancer.

The trial will test three dose levels. At each dose, the patients will receive three successive administrations, two weeks apart, NKR-2 cells. The study will enroll up to 36 patients (dose escalation and expansion phases).

ELIGIBILITY:
Inclusion Criteria:

1. Men or women ≥ 18 years old at the time of signing the ICF
2. Patients with histologically proven colorectal adenocarcinoma with potentially resectable liver metastases,
3. No previous chemotherapy for metastatic CRC,
4. The patient is due to receive first-line metastatic chemotherapy regimen with FOLFOX as a neoadjuvant
5. The patient must have an ECOG performance status 0 or 1
6. The patient must have sufficient bone marrow reserve, hepatic and renal functions

Detailed disease specific criteria exist and can be discussed with contacts listed below

Exclusion Criteria:

1. Patients who have received another cancer therapy within 2 weeks before the planned day for the apheresis
2. Patients who receive or are planned to receive any other investigational product within the 3 weeks before the planned day for the first NKR-2 administration
3. Patients who are planned to receive concurrent growth factor, systemic steroid or other immunosuppressive therapy or cytotoxic agent, other than the treatment authorized per protocol
4. Patients who underwent major surgery within 4 weeks before the planned day for the first treatment
5. Patients with uncontrolled intercurrent illness or serious uncontrolled medical disorder
6. Patients who have received a live vaccine within 6 weeks prior to the planned day for the first NKR 2 administration
7. Patients with a family history of congenital or hereditary immunodeficiency
8. Patients with history of any autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-08-07 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
The occurrence of Dose Limiting Toxicities (DLT) in all patients during the study treatment until 14 days after the first NKR-2 study treatment administration | up to resection (up to day 99 to day 126)
  DLT refers to any Grade 3 or higher toxicity or any Grade 2 or higher autoimmune toxicity that is experienced during treatment and within 14 days following the first NKR-2 dose, is new and at least possibly related to NKR-2 study treatment administered concurrently with chemotherapy
The objective response rate (ORR) before resection as measured by RECIST (version 1.1) | up to resection (up to day 99 to day 126)
  The objective response rate (ORR) is defined as the sum of the proportions of patients achieving CR or PR. The occurrence of ORR before resection will be reported.

SECONDARY OUTCOMES:
The occurrence of AEs and SAEs and any toxicity corresponding to DLT definition during the study treatment until resection visit | up to resection (up to day 99 to day 126)
  The occurrence of AEs and SAEs and any toxicity corresponding to DLT definition during the study treatment until resection visit
The occurrence of surgery complications and the wound healing status until 60 days after resection visit | until 60 days after resection
  Surgery and wound healing complications experienced within the 60-day post-operative period in patients who underwent surgery will be reported as safety endpoints
The clinical benefit rate (CBR) before resection | up to resection (up to day 99 to day 126)
  The clinical benefit rate (CBR) is defined as the proportion of patients achieving CR, PR or SD. The occurrence of CBR before resection will be reported.
The occurrence of mixed response (MR) before resection | up to resection (up to day 99 to day 126)
  The different types of MR are defined according to the following criteria: at least 30% decrease in the longest diameter (or shortest diameter for nodal lesions) occurring in at least one target lesion recorded and measured at baseline (such response occurring in otherwise SD or PD status of the sum of diameters of target lesions and without the appearance of one or more new lesions will be classified as "MR (SD)", which corresponds to a SD with target lesion regression or "MR (PD)", which corresponds to PD with target lesion regression) and the appearance of new lesion(s) in otherwise PR status of the sum of diameters of target lesions will be classified as "MR (PR)".
The resection rate | resection (day 99 to day 126)
  The presence of residual tumor following surgical resection will be assessed.
The occurrence of pathological response at surgery | resection (day 99 to day 126)
  Resected specimens. will be graded according to the two grading systems by Rubbia-Brandt et al. and Blazer et al.
The disease-free survival (DFS) or progression-free survival (PFS) | through study completion (up to month 28)
  The disease-free survival (DFS) is defined as the time from resection of liver metastases to recurrence of tumor or death from any cause. The progression-free survival (PFS) is defined as time from study registration in the study to the disease progression or death from any cause.
The event-free survival (EFS) | through study completion (up to month 28)
  The event-free survival (EFS) is defined as the time from registration in the study to any of the following events: progression, non-resectability, local or distant recurrence, or death from any cause.
The overall survival (OS) | through study completion (up to month 28)
  The overall survival (OS) is defined as the time from study registration in the study to death. If death does not occur before the patient's last study visit, then the survival will be censored at the date when patient is known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Lehmann, MD, Principal Investigator — Celyad Oncology SA
Locations (4):
- Belgium (4):
  - Institut Jules Bordet, Brussels
  - Cliniques universitaires Saint-Luc, Brussels
  - Grand Hôpital de Charleroi, Charleroi
  - UZ Leuven, Leuven

IPD SHARING:
Plan to Share IPD: No